CLINICAL TRIAL: NCT01221480
Title: Beta-Blockers Reduce Mortality and Exacerbations When Added to Stepwise Inhaled Therapy for COPD Without Adverse Effects on Lung Function.
Brief Title: What Influences Patient Outcome in Obstructive Airway Disease?
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: SHO002
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Beta Blocker Use
- No beta blocker use

SUMMARY:
The aim of this observational study is to utilise the established record linkage data available in Tayside to investigate hospital admissions, exacerbations and mortality in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Data collected through TARDIS database

Exclusion Criteria:

* History of asthma or malignancy. Less than 50 years of age

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients within NHS Tayside, UK
Sampling Method: Probability Sample
Enrollment: 5977 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality | 3000 days
  All-cause Mortality

SECONDARY OUTCOMES:
Hospital Admissions | 3000 days
  Hospital Admissions
COPD exacerbations | 3000 days
  COPD exacerbations

REFERENCES:
- [Result] Short PM, Lipworth SI, Elder DH, Schembri S, Lipworth BJ. Effect of beta blockers in treatment of chronic obstructive pulmonary disease: a retrospective cohort study. BMJ. 2011 May 10;342:d2549. doi: 10.1136/bmj.d2549. PMID 21558357